CLINICAL TRIAL: NCT06277635
Title: Effect of Silymarin Against Methotrexate-induced Liver Injury in Rheumatic Diseases, a Double-blind Randomized Controlled Trial
Brief Title: Effect of Silymarin Against Methotrexate-induced Liver Injury in Rheumatic Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAPAC001
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Psoriasis
Keywords: Rheumatoid arthritis; Psoriatric arthritis; Psoriasis; Methotrexate; Silymarin
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Psoriasis | interventions — Silymarin; milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silymarin group (Active Comparator): Silymarin 140 mg oral tid pc + methotrexate weekly + folic acid 5 mg oral OD pc for 12 weeks
  Interventions: Drug: Silymarin
- Placebo group (Placebo Comparator): Placebo + methotrexate weekly + folic acid 5 mg oral OD pc for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin — Silymarin is randomly assigned to the participants for 12 weeks during study.
  Other Names: Milk Thistle
  Arms: Silymarin group
Drug: Placebo — Placebo is randomly assigned to the participants for 12 weeks during study.
  Arms: Placebo group

SUMMARY:
To study the effect of silymarin against methotrexate-induced liver injury in rheumatic diseases including rheumatoid arthritis, psoriatric arthritis and psoriasis

DETAILED DESCRIPTION:
- Methotrexate was indeed a common and effective treatment for rheumatoid arthritis, psoriatic arthritis and psoriasis. Methotrexate-related hepatotoxicity are common occur 1:1,100 persons. Liver abnormalities varies from asymptomatic liver enzyme elevation to fatal hepatic necrosis and liver fibrosis. Methotrexate was discontinued owing to liver dysfunction in 7.4%

ELIGIBILITY:
Inclusion Criteria:

* Aged > 20 years
* Diagnosis at least one of the following

  1. Rheumatoid arthritis according to American College of Rheumatology/ The European Alliance of Associations for Rheumatology 2010(ACR/EULAR2010) with at least one joint swelling or tenderness or
  2. Psoriatric arthritis according to CASPAR classification criteria with at least one joint swelling or tenderness, or at least one site dactylitis or enthesitis or Psoriasis by dermatologist with active skin lesion
  3. No previous treatment with methotrexate or treatment with methotrexate within 30 day before randomization
  4. No previous treatment with other conventional synthetic DMARDs other than methotrexate such as sulfasalazine, hydroxycholoquine, leflunomide
  5. No previous treatment with biologic DMARDs such as anti-TNF
  6. Can follow the treatment protocal

Exclusion Criteria:

* Pregnancy or planning for pregnancy
* Breastfeeding women
* Ongoing treatment with active malignancy
* GFR < 30 ml/min/1.73m2
* Previous documented of HIV infection
* Chronic alcohol drinking ≥ 3 times/wk or drug abuse within 6 months prior to randomization
* Positive of HbsAg, anti HCV
* Previous documented of preexisting liver disease such as alcoholic liver disease, liver cirrhosis, autoimmune hepatitis
* AST or ALT > ULN ( 0-50 U/L )
* WBC < 3,000/ul or platelet < 100,000 /ul, ANC < 1,500/ul
* ILD diagnosed by rheumatologist and pulmonologist from chest X ray and HRCT
* History documented silymarin hypersensitivity or severe adverse effects diagnosed by physician or pharmacist from PMK hospital or from history drug allergy or symptoms such as rash, chest tightness, dyspnea, diarrhea and hypotension
* Cannot follow up on treatment protocal

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
AST or ALT > 1X ULN ( normal AST and ALT 0-50 U/L) | 12 weeks
  elevation of AST or ALT more than 1X ULN (% participant)

SECONDARY OUTCOMES:
AST or ALT > 2X ULN ( normal AST and ALT 0-50 U/L) AST or ALT > 2X ULN AST or ALT > 2X ULN | 12 weeks
  elevation of AST or ALT more than 2X ULN (% participant)
AST or ALT > 3X ULN ( normal AST and ALT 0-50 U/L) | 12 weeks
  elevation of AST or ALT more than 3X ULN (% participant)
AST or ALT > 5X ULN or >3X ULN ( normal AST and ALT 0-50 U/L) with symptom of hepatitis such as Fatique, abdominal pain, nausea, vomiting or total bilirubin > 2X with jaundice | 12 weeks
  elevation of AST or ALT > 5X ULN or >3X ULN with symptom of hepatitis such as Fatique, abdominal pain, nausea, vomiting or total bilirubin > 2X with jaundice (% participant)
Discontinuation rate of methotrexate | 12 weeks
  Rate of methotrexate discontinuation (%)
Adverse events | 12 weeks
  Rate of any adverse events (%)
Change of DAS-28 ESR or CRP Score | 12 weeks
  Change of DAS-28 ESR or CRP Score for patients with Rheumatoid arthritis and psoriatric arthritis (unit)
Change of BASDAI Score | 12 weeks
  Change of BASDAI Score for AS (unit)
Change of ASDAS ESR or CRP Score | 12 weeks
  Change of ASDAS ESR or CRP Score for AS (unit)
Change of BSA for psoriasis | 12 weeks
  Change of BSA for psoriasis (unit)

CONTACTS AND LOCATIONS:
Overall Officials: Rattapol Pakchotanon, M.D., Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Rheumatic Disease Unit, Department of Internal Medicine, Phramongkutklao Hospital and College of Medicine, Bangkok, Thailand, 10400, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol is to be shared with others. Full data would become available by mid 2026.
Supporting Information: Study Protocol
Time Frame: mid 2026
Access Criteria: IPD Sharing Access Criteria has not been decided.